CLINICAL TRIAL: NCT01103089
Title: Observations From Long Term Responders in the Gefitinib (Iressa) Expanded Access Program (EAP)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-ONL-IRE-2009/1
Record Dates: First submitted 2010-04-05; First posted 2010-04-14 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; EGFR; gefitinib; observational
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to determine patient characteristics from patients that have used Iressa for a period of minimal 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the gefitinib Expanded Access Program
* Patient still uses gefitinib in September 2009

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the gefitinib Expanded Access Programme in the Netherlands.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The following characteristics of the 'long-term responders' from the EAP; gender, ethnicity, smoking history (pack years), EGFR-TK mutation and histology of NSCLC. | Characteristics will be recorded once, retrospectively

SECONDARY OUTCOMES:
To assess the long-term safety in subjects treated with gefitinib by collecting information on: All adverse events that have lead to an interruption/reduction of gefitinib or another intervention | Once, retrospectively for the period the patient has used gefitinib (minimal 3 years)
long-term safety in subjects; what real life data measures are being taken by lung physicians to counter side effects caused by long term gefitinib treatment; the number, reason, effect and description of interventions that have been taken | Once, retrospectively for the period the patient has used gefitinib (minimal 3 years)
long-term safety: Number, reason and effect of interruptions during gefitinib use to determine side effects typical for the long-term treatment with gefitinib | Once, retrospectively for the period the patient has used gefitinib (minimal 3 years)

CONTACTS AND LOCATIONS:
Locations (11):
- Netherlands (11):
  - Research Site, Amsterdam
  - Research Site, Apeldoorn
  - Research Site, Groningen
  - Research Site, Helmond
  - Research Site, Hengelo
  - Research Site, Hoofddorp
  - Research Site, Leiden
  - Research Site, The Hague
  - Research Site, Veldhoven
  - Research Site, Venlo
  - Research Site, Zutphen